CLINICAL TRIAL: NCT05885308
Title: Intervening for Increased Quality of Life Among Older People in Sweden
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karlstad University (Other)
Responsible Party: Principal Investigator, Johanna Gustavsson, Lecturer, Karlstad University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20210102
Record Dates: First submitted 2023-05-12; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Physical Inactivity; Mental Health Issue
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group training (Active Comparator)
  Interventions: Behavioral: Otago
- Online training (Experimental)
  Interventions: Behavioral: Otago

INTERVENTIONS:
Behavioral: Otago — Group training is compared with training performed at participants' homes, using an online film

SUMMARY:
In the wake of the Covid-19 pandemic, Sweden and other countries have become aware of how life has changed; the world is now a "hybrid world" where many daily activities have moved online. The forced physical isolation has also led to an increase in depression and loneliness, especially among elderly people. Traditional interventions often involve physical contact, and there are valuable lessons to be learned from this situation, where physical isolation is forced, in order to mitigate the consequences both during and after this pandemic.

The overall purpose of this project is to study physical activity as a way to engage in and maintain an active lifestyle and /or increase the quality of life and limit mental health problems for older people and to study how scalability, accessibility, commitment, and adherence can be improved with flexible programs with digital tools. The specific research question is:

Is there a difference between the online exercise program and the onsite exercise program in terms of physical activity, balance, motivation, quality of life and mental health?

The results are expected to give insights into how to increase physical activity using flexible programs with digital options and to maintain quality of life among the elderly. By giving the elderly population different options for being physically active and thereby empowering this group, this project contributes to creating a socially sustainable community in which elderly citizens are included.

ELIGIBILITY:
Inclusion Criteria:

* Understand Swedish

Exclusion Criteria:

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity | Time points: 0, 3 and 6 months
  The International Physical Activity Questionnaire (IPAQ) (for older people) measures physical activity where the individual self-reports the number of minutes spent inactive and active (Sember et al., 2020).
  The number of steps will be measured with a pedometer.
Change in leg strength and endurance | Time points: 0, 3 and 6 months
  30-Second Chair Stand will be used to test leg strength and endurance (Jones et al 2000). The investigator record the number of times the patient stands in 30 seconds. A below average score indicates a risk for falls. For example, a below average score for men aged 70-74 is < 12 and < 10 for women.

SECONDARY OUTCOMES:
Change in depression | Time points: 0, 3 and 6 months
  GDS 20 (Geriatric Depression Scale) is a screening instrument with 20 items to identify depression in older people (Brink, T. L. et al 1982). The questions are answered with yes or no, and answers indicating issues (sometimes yes, sometimes no) are given one point. Scores of 0-5 on the scale are interpreted as depression being unlikely, while scores of 6-20 are interpreted as possible suspicion of depression.
Change in Quality Of Life | Time points: 0, 3 and 6 months
  EQ-5D-5L measures Quality Of Life and comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The maximum score of 1 indicates the best health state In addition, the individual self-report their health on a scale from 0-100, where 100 represented the best health (https://euroqol.org/eq-5d-instruments/eq-5d-5l-about/; Burström et al., 2020; Feng, Kohlmann, Janssen, & Buchholz, 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Gustavsson, PhD, Principal Investigator — Karlstad University
Locations (1):
- Karlstad University, Karlstad, Värmland County, Sweden

IPD SHARING:
Plan to Share IPD: No